CLINICAL TRIAL: NCT04638959
Title: Faecal Bacteria Detection in Early Screening and Diagnosis of Gastric Cancer: a Large-scale Multi-center Case-control Study
Brief Title: Study of Faecal Bacteria Detection in Early Screening and Diagnosis of GC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai Changzheng Hospital (Other); Ruijin Hospital (Other); Jing'an District Central Hospital of Shanghai (Unknown); Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other); Nanfang Hospital, Southern Medical University (Other); Seventh Medical Center of PLA Army General Hospital (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Zhongshan Hospital Xiamen University (Other); Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Jing-yuan Fang, MD, Ph. D, Professor, Shanghai Jiao Tong University School of Medicine
Other Study IDs: KY[2019]130
Record Dates: First submitted 2020-11-18; First posted 2020-11-20 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Non-invasive and Sensitive Faecal Bacterial Markers for Early Screening and Diagnosis of Gastric Cancer
Keywords: faecal bacterial marker; early screening and diagnosis; gastric cancer
MeSH Terms: conditions — Disease; Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — gastric cancer tissues gastric mucosa stools
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GC: patients diagnosed with GC
  Interventions: Other: collect gastric tissue and stool samples
- HC: patients diagnosed with chronic gastritis by histopathology
  Interventions: Other: collect gastric tissue and stool samples

INTERVENTIONS:
Other: collect gastric tissue and stool samples — collect gastric tissue and stool samples

SUMMARY:
In this clinical trial, we aim to explore the synergistic alteration of specific bacteria both in gastric mucosas and feces of gastric cancer patients for the method of non-invasive and cost-effective faecal marker detection. We aim to select and validate specific microbes as noninvasive, accurate, simple, sensitive and highly-accepted biomarkers that might assist to screen and diagnose gastric cancer, especially early gastric cancer patients.

DETAILED DESCRIPTION:
We conducted a large-scale multi-centre retrospective case-control study. Approximately a total of 1080 volunteers aging 40-75 in three independent cohorts, discovery cohort, validation cohort 1, validation cohort 2, will be recruited from 10 hospitals throughout China. Among them, 530 subjects in both discovery cohort and validation cohort 1 were from Shanghai Jiao Tong University School of Medicine Renji Hospital from August to December in 2018. Around 550 participants will be enrolled in validation cohort 2 from nine hospitals in China.Each cohort recruits both patients diagnosed with GC (GC group) and gender, age and body mass index (BMI)-matched healthy-control (HC) individuals diagnosed with chronic gastritis by histopathology). Individuals enrolled were either asymptomatic undergoing upper GI endoscopy screening or went to GI clinic with digestive symptoms. Subjects in HC group are conducted colonoscopy within 0.5 year before or after upper endoscopy. We collect gastric tissue biopsies and stool samples from gastric cancer patients and healthy-controls. First in the discovery cohort, which will recruit 20 subjects, 13 pairs of both cancerous & noncancerous gastric tissues and pre-operation feces in GC group will be collected. 7 subjects provide their paired mucosal biopsies and stools in HC group before examination. 16S ribosomal RNA gene sequencing will be used to select the synergistically differential bacteria species as well as find out microbial compositional distinction and diversity from both tissue and stool samples between GC and HC group. Second, the validation cohort 1 recruiting a total of 510 subjects (294 GC patients and 216 HC individuals), 217 pre-operation faecal specimens and 141 fresh tissues (cancerous & noncancerous tissues) from GC group, and 127 faecal samples and 124 gastric biopsies will be collected. Quantitative PCR (qPCR) will be used to validate the high-throughput sequencing results in discovery cohort in a single center. Among them, 35 objects in HC group and 64 patients in GC group will provide their paired tissues and feces. Third, in validation cohort 2, we are going to enroll volunteers from multiple geographic locations to confirm our results. 550 stool samples will be collected to further validate the accuracy, sensitivity and specificity of the cut-off value analyzed from validation cohort 1. All results of laboratory tests including tumor markers CEA, CA199,CA724 were obtained from the electronic query system. The GC stages will be assessed by the TNM system according to AJCC Version 4.2017 based on surgical records, histopathology and radiographic images (eg. PET-CT, abdominal enhanced CT). All subjects will sign up informed consent form before sample collection. The protocol of present study was approved by Ethics Review Committee of all participating hospitals.

ELIGIBILITY:
Inclusion Criteria:

* 1）Age between 40 and 75;
* 2）Subjects in GC group are pathologically diagnosed as gastric cancer prior to any treatment such as surgery, endoscopic resection, chemotherapy, radiotherapy, immunotherapy, traditional Chinese medicine therapy, etc. The results of their preoperative abdominal enhanced CT or PET-CT indicated no obvious bowel abnormalities (inflammation, polyps, ulcers, tumors, erosions, melanosis, etc.);
* 3) Subjects in HC group are diagnosed with chronic gastritis by endoscopy and pathology. without ulcers, polyps, tumors, severe erosions or bile reflux, and no obvious abnormal findings (inflammation, polyps, ulcers, tumors, erosions, melanosis, etc.) by colonoscopy within half a year;
* 4) Subjects are willing to cooperate with this research and provide stool/mucosa samples as required.

Exclusion Criteria:

* 1) with severe systemic infection, nasopharyngeal/oral cavity inflammation (periodontitis, gingivitis, tonsillitis, etc.), respiratory tract infection, soft tissue or skin infection, abscess or endocarditis within 3 months prior to recruitment;
* 2）prior medication history of the following medicine within 3 months: nonsteroidal anti-inflammatory drugs (NSAIDs), immunosuppressor, antibiotics, probiotics, hormones or immune-suppressants at least 1 week;
* 3）prior medication history of proton-pump inhibitors or H2 receptor inhibitors for over 2 months within 1 year;
* 4) with a history of H.pylori eradication therapy within 1 year;
* 5) with severe constipation, diarrhea or defecation habits changes within 3 months;
* 6) personal history of cancer, organ transplantation, parasites infection or other severe digestive system diseases (inflammatory bowel disease, liver cirrhosis, etc.);
* 7) with uncontrolled digestive bleeding, obstruction, perforation and any trauma or surgery within 3 months;
* 8) with uncontrolled chronic metabolic or endocrine disorders, e.g. hypertension, diabetes, hyperlipidemia, hyperuricemia, etc.
* 9) on a vegetarian diet or with great changes of eating habits within 3 months;
* 10) refusal of participate in this study.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants are required to complete a structured questionnaire for assessment of inclusion requirement.
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2019-09-30 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
differences in abundance of gut microbiota | 1 year
  differences in abundance of gut microbiota for participants with different clinical outcomes confirmed by qPCR(quantitive polymerase chain reaction)

SECONDARY OUTCOMES:
evidence of gastric carcinoma | 1 year
  Different outcomes for gastric carcinoma confirmed by endoscopy and pathology

OTHER OUTCOMES:
Basic information of patients with different clinical outcomes | 1 year
  Basic information of patients with different clinical outcomes by a questionnaire

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - Department of Gastroenterology, the Seventh Medical Center of PLA General Hospital, Beijing, Beijing Municipality
  - Department of Gastroenterology, Zhongshan Hospital, Xiamen University, Xiamen, Fujian
  - Department of Gastroenterology, Nanfang Hospital, Southern Medical Univerisity, Guangdong, Guangzhou
  - Division of Gastroenterology and Hepatology, The Affiliated DrumTower of Nanjing University Medical School, Nanjing, Jiangsu
  - Division of Gastroenterology and Hepatology, Ren-Ji Hospital, Shanghai Jiao-Tong University School of Medicine, Shanghai Institute of Digestive Disease; Key Laboratory of Gastroenterology & Hepatology, Ministry of Health, Shanghai, Shanghai Municipality
  - Department of Gastroenterology and Hepatology, General Hospital, Tianjin Medical University, Tianjin, Tianjin Municipality
  - Jing'an District Central Hospital of Shanghai, Shanghai
  - Shanghai Changzheng Hospital, Shanghai
  - Shanghai Ninth People's Hospital, Shanghai
  - Shanghai Ruijin Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhou CB, Pan SY, Jin P, Deng JW, Xue JH, Ma XY, Xie YH, Cao H, Liu Q, Xie WF, Zou XP, Sheng JQ, Wang BM, Wang H, Ren JL, Liu SD, Sun YW, Meng XJ, Zhao G, Chen JX, Cui Y, Wang PQ, Guo HM, Yang L, Chen X, Ding J, Yang XN, Wang XK, Qian AH, Hou LD, Wang Z, Chen YX, Fang JY. Fecal Signatures of Streptococcus anginosus and Streptococcus constellatus for Noninvasive Screening and Early Warning of Gastric Cancer. Gastroenterology. 2022 Jun;162(7):1933-1947.e18. doi: 10.1053/j.gastro.2022.02.015. Epub 2022 Feb 12. PMID 35167866